CLINICAL TRIAL: NCT06280144
Title: Multi-center, Randomized, Double-blind, Placebo-controlled Trial of a Live Attenuated Influenza Vaccine in People Aged 3-17
Brief Title: Post-marketing Study of Lyophilized Nasal Spray Live Attenuated Influenza Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Collaborators: Hu Bei province Center for Disease control and prevention (Unknown); The Inner Mongolia Autonomous Region Center for Disease Control and Prevention (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PF20230428
Record Dates: First submitted 2023-09-01; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2023-12

CONDITIONS: Influenza Prevention
Keywords: Protection effect
MeSH Terms: interventions — Influenza Vaccines; Freeze Drying; Inhalation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Influenza Vaccine, Live, Nasal, Freeze-dried
  Interventions: Biological: Influenza Vaccine, Live, Nasal, Freeze-dried
- Placebo group (Placebo Comparator): Sterile water for inhalation
  Interventions: Other: Sterile water for inhalation

INTERVENTIONS:
Biological: Influenza Vaccine, Live, Nasal, Freeze-dried — The titer of live attenuated influenza virus containing A (H1N1) and A (H3N2) should not be less than 6.9 lg EID50, and the titer of live attenuated influenza B virus should not be less than 6.4 lg EID50
  Arms: Experimental group
Other: Sterile water for inhalation — Sterile water for inhalation
  Arms: Placebo group

SUMMARY:
To evaluate the protective effect 14 days after the live attenuated influenza vaccine; To evaluate the protective effect of vaccination with live attenuated influenza vaccine; To evaluate the safety of freeze-dried nasal spray live attenuated influenza vaccine; To evaluate the detoxification and genetic stability of lyophilized nasal spray vaccine.

To evaluate the protective effect of novel coronavirus after 14 days of inoculation with the live attenuated influenza vaccine.

DETAILED DESCRIPTION:
Main end point:

Primary influenza protective effect endpoint Protective effect of 14 days on laboratory-confirmed influenza cases. Protective effect of 14 days after receiving lyophilized nasal spray live attenuated influenza vaccine on laboratory-confirmed serotype influenza cases.

Secondary endpoints:

Secondary point of secondary endpoint Protective effect of freeze-dried nasal spray live attenuated influenza vaccine 0 days later on laboratory-confirmed influenza cases.

Protective effect of freeze-dried nasal spray live attenuated influenza vaccine 14 days later on clinically diagnosed influenza cases.

Protective effect of live attenuated influenza-like vaccine 14 days against influenza-like cases.

safety Incidence of adverse events and serious adverse events within 0-30 days after immunization.

Study on detoxification Proproportion of vaccine attenuated proportion and vaccine attenuated content (titer) at different times after vaccination (days 3,7,15).

Exploration endpoint:

14 days after the freeze-dried nose vaccine, the vaccine was protective for the detection of COVID-19 cases.

ELIGIBILITY:
Inclusion Criteria:

1. Local residents aged between 3 and 17;
2. People who signed the informed consent form and could actively cooperate with the study；
3. Axillary body temperature of 37.0℃.

Exclusion Criteria:

1. Subjects who meet the contraindications and precautions specified in the vaccine instructions:

   1. Those known to be allergic to any ingredients of this product, including eggs, excipients, gentamycin sulfate;
   2. Patients with acute disease, severe chronic disease, the acute onset of chronic disease and fever;
   3. Women in pregnancy;
   4. Patients with Leigh syndrome treated with aspirin or aspirin-containing drugs;
   5. Immunodeficient, immunocompromised, or under immunosuppressive therapy;
   6. Patients with uncontrolled epilepsy and other progressive neurological diseases, patients with a history of Guillain-Barre syndrome; And g. patients with rhinitis (with a clear diagnosis and in the onset of rhinitis).
2. Have received other clinical study drugs or were participating in other clinical trials within 1 month before entering the cohort.
3. Have received any influenza vaccine during this natural year before entering the study
4. Those who have been diagnosed with influenza in this natural year before entering the study.
5. Any condition that the investigator judged to affect the trial.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 6080 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Primary influenza protective effect endpoint | 7 months
  Protective effect of freeze-dried nasal spray live attenuated influenza vaccine 14 days on the incidence of laboratory-confirmed influenza cases
Primary influenza protective effect endpoint | 7 months
  Protective effect of 14-day live attenuated influenza vaccine on the incidence of laboratory-confirmed cases of serotype influenza.

SECONDARY OUTCOMES:
Secondary protective efficacy endpoint | Seven months
  Protective effect of freeze-dried nasal spray live attenuated influenza vaccine after 0 days on the incidence of laboratory-confirmed influenza cases.
Secondary protective efficacy endpoint | Seven months
  Protective effect of freeze-dried nasal spray live attenuated influenza vaccine 14 days later on the incidence of clinically diagnosed influenza cases.
Secondary protective efficacy endpoint | Seven months
  Protective effect of 14 days on the incidence of influenza-like cases.
Safety | One month
  Incidence of adverse events and serious adverse events within 0-30 days .AE at the inoculation site: runny nose / nasal congestion, sore throat Non-inoculation site (systemic) AEs (including vital signs): fever, cough, headache, fatigue, fatigue, nausea, vomiting, muscle pain, arthralgia, chills, anorexia, acute anaphylaxis (type I hypersensitivity).
  Other AEs, SAEs, and pregnancy events incidence.
Study on detoxification | 15 days
  Proproportion of vaccine attenuated proportion and vaccine attenuated content (titer) at different times after vaccination (days 3,7,15).

OTHER OUTCOMES:
Protective effect of COVID-19 cases. | Seven months
  14 days after inoculation of freeze-dried nasal influenza vaccine, the vaccine protected the incidence of COVID-19 cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Chifeng, Inner Mongolia, China

IPD SHARING:
Plan to Share IPD: Undecided